CLINICAL TRIAL: NCT04692818
Title: 3D Multimodal Ultrasound Imaging for Breast Cancer
Brief Title: 3D Ultrasound Breast Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-010751; W81XWH-21-1-0063 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Breast Tumor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Clinically indicated breast tumor biopsy (Experimental): Subjects with breast lesion and are scheduled for clinically-indicated biopsy will have 3D Multimodal Ultrasound Imaging performed
  Interventions: Diagnostic Test: GE Logiq E10 clinical ultrasound scanner; Diagnostic Test: Verasonics research scanner

INTERVENTIONS:
Diagnostic Test: GE Logiq E10 clinical ultrasound scanner — 2D B-mode, Doppler, and shear wave elastography images of the lesion
Diagnostic Test: Verasonics research scanner — 3D B-mode imaging, microvessel imaging, and shear wave elastography

SUMMARY:
The purpose of this research is to study the efficacy of a new ultrasound imaging method for diagnosis of breast mass.

ELIGIBILITY:
Inclusion Criteria:

* Adult women ≥ 18 years of age.
* solid breast lesion and ultrasound guided biopsy (either as part of their clinical care or through participation in other IRB-approved studies)
* lesion size of 3mm or larger

Exclusion Criteria:

* < 18 years of age.
* Lacking capacity to consent
* Pregnant or lactating
* Receiving cancer therapy such as chemotherapy or radiation therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
BI-RADS Score | Baseline
  BI-RADS scores will be obtained using 2D B-mode ultrasound images from the GE Logiq E10 clinical scanner, and using 3D B-mode images from the Verasonics scanner. A 7-point BI-RADS scale will be used, with a score of 1, 2, or 3 considered negative and 4a, 4b, 4c, and 5 considered positive.

CONTACTS AND LOCATIONS:
Overall Officials: Shigao Chen, PhD, Principal Investigator — Mayo Clinic; Christine Lee, MD, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials